CLINICAL TRIAL: NCT01593384
Title: To Determine the Clinical Impact of the Combination of Digital Breast Tomosynthesis and Digital Mammography on Screening for Breast Cancer
Brief Title: Prospective Chart-Review: Impact of Combination - Digital Breast Tomosynthesis + Digital Mammography
Status: Withdrawn | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE2112
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Digital Breast Tomosynthesis (DBT); Digital Mammography (DM)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Digital Breast Tomosynthesis (DBT) is a technology that has been developed to improve lesion detection in dense breasted women. Even though DBT has been regarded as a study for dense breasted women, it may also improve lesion detection at an earlier stage and smaller size in women with less dense breast tissue. The overlapping of tissue on a standard of care 2D mammogram leads to decreased cancer detection, it also contributes to pseudo lesions that mimic cancers. This leads to patients being asked to come back for additional imaging including mammogram and/or ultrasound images. DBT has shown to decrease call back rates by up to 43% in reader studies. Even though these results are promising they were not done in a realistic clinical setting.The purpose of this study is to evaluate the FDA-approved combination standard digital mammography (DM) and DBT technology and its impact on our clinical practice.

DETAILED DESCRIPTION:
The investigators would like to prospectively measure the impact on recall rates, comparing DM (digital mammography) and DM+DBT, in our practice and the impact on cancer detection in our screening population. This is a two-site study in which all asymptomatic subjects undergoing the FDA-approved combination standard of care Digital Mammogram and Digital Breast Tomosynthesis (DM+DBT) exam will be eligible for the trial. Each subject will be her own control.Only radiologists who have gone through 8 hours of Tomosynthesis training will interpret the DM and DBT images. These radiologists will categorize each case as either dense (BI-RADS density score of 3 or 4) or fatty (BI-RADS density score of 1 or 2). The radiologist will initially read the standard of care DM part of the study first and record their interpretation and final BIRADs category. The same radiologist will then interpret the DM+DBT combination study and record their final interpretation and BIRADs category. Prior mammogram studies will be used for comparison when reading the DM and DM+DBT studies.

ELIGIBILITY:
Inclusion Criteria:

* Female ages 30 and over
* Asymptomatic
* Any ethnic origin
* No contraindication for routine bilateral mammogram

Exclusion Criteria:

* Pregnancy
* Lactating patients
* Breast implants
* Unable to understand and execute written informed consent
* Patient unable to obtain a mammogram while standing without assistance

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from routine clinical patient population at our medical facility. There will be inclusion of employees and students in the study. A number of UHCMC employees and a few CWRU students are in our routine clinical patient population.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Measure the impact on recall rates, comparing DM and DM+DBT | 3 yrs
  Measure the impact on recall rates, comparing DM and DM+DBT, in our practice and the impact on cancer detection in our screening population.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Plecha, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center